CLINICAL TRIAL: NCT01211483
Title: Randomized, Placebo-controlled, Double-blind Phase 1b/2 Study of U3-1287 (AMG 888) in Combination With Erlotinib in EGFR Treatment Naïve Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC) Who Have Progressed on at Least One Prior Chemotherapy
Brief Title: Study of Erlotinib With or Without Investigational Drug (U3-1287) in Subjects With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U31287-A-U201
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — patritumab; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A: U3-1287 (high dose) + Erlotinib (Experimental): U3-1287 (high dose) intravenously (IV) every three weeks (Q3W) + Erlotinib 150 mg/day orally (PO) until cancer gets worse, side effects become unacceptable or participant withdraws consent
  Interventions: Drug: U3-1287; Drug: Erlotinib
- Part B: U3-1287 (low dose) + Erlotinib (Experimental): U3-1287 (low dose) IV Q3W + Erlotinib 150 mg/day PO until cancer gets worse, side effects become unacceptable or participant withdraws consent
  Interventions: Drug: U3-1287; Drug: Erlotinib
- Part B: Placebo + Erlotinib (Placebo Comparator): Placebo matching U3-1287 IV Q3W + Erlotinib150 mg/day PO until cancer gets worse, side effects become unacceptable or participant withdraws consent
  Interventions: Drug: Erlotinib; Drug: Placebo

INTERVENTIONS:
Drug: U3-1287 — Liquid 70 mg/mL for IV infusion at high dose or low dose
  Other Names: Patritumab
  Arms: Part A: U3-1287 (high dose) + Erlotinib; Part B: U3-1287 (low dose) + Erlotinib
Drug: Erlotinib — Tablet 150 mg for oral administration
Drug: Placebo — Placebo liquid matching U3-1287 for IV infusion
  Arms: Part B: Placebo + Erlotinib

SUMMARY:
This is a Phase 1b/2 study. In Phase 1b, subjects will know the treatment they are receiving. Subjects will receive Erlotinib + U3-1287. The Phase 1b portion will determine if adding U3-1287 to Erlotinib will be safe in subjects with advanced non-small cell lung cancer who fail prior treatment. In the Phase 2 portion, subjects will be blinded to the treatments they are receiving. Subjects will receive either Erlotinib alone or Erlotinib + U3-1287.

The Phase 2 portion will determine if adding U3-1287 to Erlotinib will be safe and improve survival in subjects with advanced non-small cell lung cancer who failed the first treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Histologically or cytologically confirmed stage IIIB not amenable to surgery or curative intent or stage IV NSCLC.
* Disease progression or recurrence following treatment after last chemotherapy or chemoradiation regimen (completed within the previous 12 months) documented by radiographic assessment.
* Measurable disease by Response Evaluation Criteria for Solid Tumors v1.1 (RECIST v1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone marrow, renal, and hepatic function.
* Prothrombin time and partial thromboplastin time ≤1.5 x upper limit of normal (ULN).
* Availability of recent (before treatment start) or archival tumor specimens (Phase 2 participants only).
* For female participants, must be postmenopausal, surgically sterile, or must use maximally effective birth control during the period of therapy, and must be willing to use effective contraception up to 6 months after the last dose of study drug and had a negative urine or serum pregnancy test before entry into the study if female participants were of childbearing potential.
* For male participants, must be surgically sterile or willing to use a double barrier contraception method upon enrollment, during the course of the study, and for 6 months following the last investigational drug dose
* Written informed consent.

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 45%.
* Prior epidermal growth factor receptor (EGFR)-targeted regimen, anti-HER2, anti-HER3, or anti-HER4 therapy.
* More than 2 prior chemotherapy regimens for NSCLC (Phase 2 participants only).
* History of other malignancies, except adequately treated nonmelanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years.
* History of corneal disease.
* History of interstitial lung disease.
* Clinically active brain metastases, defined as untreated symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Participants with treated brain metastases that were no longer symptomatic and required no treatment with steroids could be included in the study if they had recovered from the acute toxic effect of radiotherapy.
* Uncontrolled hypertension (diastolic > 100 mmHg or systolic > 140 mmHg).
* Clinically significant electrocardiogram changes that obscured the ability to assess the respiratory rate, pulse rate, QT, QTc, and QRS intervals.
* Ascites or pleural effusion requiring chronic medical intervention.
* Myocardial infarction within 1 year before enrollment, symptomatic congestive heart failure (New York Heart Association > Class II), unstable angina, or unstable cardiac arrhythmia requiring medication.
* Treatment with anticancer therapy, antibody based therapy, retinoid therapy, or hormonal therapy within 4 weeks before study treatment or treatment with nitrosoureas or mitomycin C within 6 weeks before study drug treatment or treatment with small molecule tyrosine kinase inhibitors (TKIs) within 2 weeks before study drug treatment. Prior and concurrent use of hormone replacement therapy was permitted.
* Therapeutic radiation or major surgery within 4 weeks before study treatment or palliative radiation therapy within 2 weeks before study drug treatment.
* Participated in clinical drug trials within 4 weeks (2 weeks for small molecule TKIs) before study drug treatment. Current participation in other investigational procedures.
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection.
* History of hypersensitivity to any of the study drugs or to any excipients.
* Concurrent use of CYP3A4 inducers or inhibitors.
* Any known pre-existing condition including substance abuse that could interfere with participant's participation in and completion of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (52):
- United States (14):
  - Glendale, Arizona
  - TRM - Oncology Research Associates, PLLC, d/b/a Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Anaheim, California
  - Encinitas, California
  - La Verne, California
  - Los Angeles, California
  - Orlando, Florida
  - Atlanta, Georgia
  - Joliet, Illinois
  - Evansville, Indiana
  - Baton Rouge, Louisiana
  - Detroit, Michigan
  - The Bronx, New York
  - York, Pennsylvania
- Austria (2):
  - Graz
  - Innsbruck
- Belgium (2):
  - Ghent
  - Liège
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Germany (10):
  - Essen
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Gauting
  - Halle
  - Hamburg
  - Herne
  - Löwenstein
  - Mainz
  - Tübingen
- Hungary (2):
  - Budapest
  - Pécs
- Israel (3):
  - Petah Tikva
  - Tel Aviv
  - Tel Litwinsky
- Italy (4):
  - Lido di Camaiore
  - Piacenza
  - Pisa
  - Reggio Emilia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Romania (2):
  - Suceava
  - Târgu Mureş
- Golnik, Slovenia
- Ukraine (6):
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Sumy
  - Uzhhorod
- United Kingdom (2):
  - London
  - Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 222 participants who met all inclusion criteria and no exclusion criteria were enrolled in this Phase 1b/Phase 2 study at 52 sites in Europe and Israel and 14 sites in the United States.
Pre-assignment Details: Of the 222 participants enrolled, 3 were randomized but not dosed. Two participants died before dosing and 1 participant withdrew the consent. Data on the 219 participants are presented in this report.
Groups:
- Phase 1b: U31287 18 mg/kg + Erlotinib: Participants who received U3-1287 18 mg/kg intravenously (IV) every three weeks (Q3W) and Erlotinib 150 mg/day orally (PO).
- Phase 2: U3-1287 18 mg/kg + Erlotinib: Participants who were randomized to receive U3-1287 18 mg/kg intravenously (IV) every three weeks (Q3W) and Erlotinib 150 mg/day orally (PO).
- Phase 2: U3-1287 9 mg/kg + Erlotinib: Participants who were randomized to receive U3-1287 9 mg/kg IV Q3W and Erlotinib 150 mg/day PO.
- Phase 2: Placebo + Erlotinib: Participants who were randomized to receive placebo matching U3-1287 IV Q3W and Erlotinib150 mg/day PO.
Period: Phase 1b
Arm/Group | Phase 1b: U31287 18 mg/kg + Erlotinib | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Started | 7 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 0
Not completed — Death | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b: U31287 18 mg/kg + Erlotinib | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Started | 0 | 72 (Participants entered only at Period 2.) | 72 (Participants entered only at Period 2.) | 71 (Participants entered only at Period 2.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 72 | 72 | 71
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2
Not completed — Death | 0 | 64 | 53 | 53
Not completed — Withdrawal by Subject | 0 | 1 | 10 | 5
Not completed — Study terminated by Sponsor | 0 | 6 | 8 | 11

BASELINE CHARACTERISTICS:
Population: Baseline and demographic characteristics are reported in patients enrolled in Phase 1b/Phase 2 of study.
Groups:
- Phase 1b: U3127 18mg/kg + Erlotinib: Participants who received U3-1287 18 mg/kg intravenously (IV) every three weeks (Q3W) and Erlotinib 150 mg/day orally (PO).
- Total: Total of all reporting groups
Arm/Group | Phase 1b: U3127 18mg/kg + Erlotinib | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib | Total
Number analyzed (Participants) | 7 | 70 | 71 | 71 | 219
Age, Continuous [Median (Full Range); unit: years] | 68 [48 to 78] | 62.0 [41 to 82] | 65.0 [44 to 84] | 60.0 [35 to 88] | 62.5 [35 to 88]
Age, Customized [Count of Participants; unit: Participants]
  <60 years | 2 | 28 | 24 | 33 | 87
  ≥60 years | 5 | 42 | 47 | 38 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 32 | 23 | 28 | 86
  Male | 4 | 38 | 48 | 43 | 133
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 7 | 68 | 71 | 69 | 215
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Progression-free survival (PFS) was defined as the time from the date of randomization to the earlier of the dates of first objective documentation of radiographic disease progression or death due to any cause (as per Response Evaluation Criteria in Solid Tumors [RECIST] Version 1.1).
Time Frame: Time from the randomization date up to the date of first objective documentation of disease progression or death due to any cause (whichever comes first), up to 3 years 2 months
Population: Progression-free survival was assessed in the Full Analysis Set in Phase 2 of the study. Efficacy was not assessed in the Phase 1b portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 70 | 71 | 71
months | 1.4 [1.3 to 2.7] | 2.5 [1.5 to 3.0] | 1.6 [1.4 to 2.6]
Statistical Analysis 1: Comparison: Phase 2: U3-1287 18 mg/kg + Erlotinib vs Phase 2: Placebo + Erlotinib; Test type: Superiority; Hazard Ratio (HR) = 0.978, 95% CI 2-sided [0.674 to 1.420]
Statistical Analysis 2: Comparison: Phase 2: U3-1287 9 mg/kg + Erlotinib vs Phase 2: Placebo + Erlotinib; Test type: Superiority; Hazard Ratio (HR) = 0.770, 95% CI 2-sided [0.523 to 1.131]

2. Primary Outcome: Progression-Free Survival in Participants With High Heregulin-Expressing Tumors Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Progression-free survival (PFS) was defined as the time from the date of randomization to the earlier of the dates of first objective documentation of radiographic disease progression or death due to any cause (as per Response Evaluation Criteria in Solid Tumors [RECIST] Version 1.1). Heregulin (HRG) high is defined as delta cycle threshold value < 3.9.
Time Frame: as for outcome 1
Population: Progression-free survival was assessed in participants with high heregulin-expressing tumors in the Full Analysis Set in Phase 2 of the study. Efficacy was not assessed in the Phase 1b portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 17 | 16 | 18
months | 3.4 [1.2 to 5.7] | 3.0 [1.5 to 5.7] | 1.4 [1.2 to 2.3]
Statistical Analysis 1: Comparison: Phase 2: U3-1287 18 mg/kg + Erlotinib vs Phase 2: Placebo + Erlotinib; Test type: Superiority; p = 0.0185, Cox proportional hazard; Hazard Ratio (HR) = 0.369, 95% CI 2-sided [0.161 to 0.846]
Statistical Analysis 2: Comparison: Phase 2: U3-1287 9 mg/kg + Erlotinib vs Phase 2: Placebo + Erlotinib; Test type: Superiority; p = 0.0034, Cox proportional hazard; Hazard Ratio (HR) = 0.288, 95% CI 2-sided [0.125 to 0.663]

3. Primary Outcome: Progression-Free Survival in Participants With Low Heregulin-Expressing Tumors Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Progression-free survival (PFS) was defined as the time from the date of randomization to the earlier of the dates of first objective documentation of radiographic disease progression or death due to any cause (as per Response Evaluation Criteria in Solid Tumors [RECIST] Version 1.1). Heregulin (HRG) low is defined as a delta cycle threshold value ≥ 3.9.
Time Frame: as for outcome 1
Population: Progression-free survival was assessed in participants with low heregulin-expressing tumors in the Full Analysis Set in Phase 2 of the study. Efficacy was not assessed in the Phase 1b portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 19 | 15 | 16
months | 1.4 [1.1 to 8.5] | 2.1 [1.3 to 3.0] | 1.4 [1.3 to 8.1]
Statistical Analysis 1: Comparison: Phase 2: U3-1287 18 mg/kg + Erlotinib vs Phase 2: Placebo + Erlotinib; Test type: Superiority; p = 0.9879, Cox proportional hazard; Hazard Ratio (HR) = 1.006, 95% CI 2-sided [0.458 to 2.212]
Statistical Analysis 2: Comparison: Phase 2: U3-1287 9 mg/kg + Erlotinib vs Phase 2: Placebo + Erlotinib; Test type: Superiority; p = 0.6276, Cox proportional hazard; Hazard Ratio (HR) = 1.222, 95% CI 2-sided [0.544 to 2.746]

4. Secondary Outcome: Overall Survival Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Overall Survival (OS) was defined as the time from the randomization date to the date of death.
Time Frame: Time from the randomization date up to the date of death due to any cause, up to 3 years 2 months
Population: Overall survival was assessed in Full Analysis Set in Phase 2 of the study. Efficacy was not assessed in the Phase 1b portion of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 70 | 71 | 71
months | 5.3 [4.0 to 6.9] | 6.3 [4.7 to 9.3] | 7.2 [5.4 to 10.6]

5. Secondary Outcome: Objective Response Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Objective response was defined as the best response of either complete response (CR) or partial response (PR). As per Response Evaluation Criteria in Solid Tumors Version 1.1, CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Time from date of randomization up to date of first documentation of objective response of either CR or PR (whichever comes first), up to 3 years 2 months
Population: Objective response rate was assessed in participants with measurable disease in the Full Analysis Set in Phase 2 of the study. Efficacy was not assessed in the Phase 1b portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 70 | 70 | 71
Participants | 6 | 9 | 4

6. Secondary Outcome: Time to Objective Response Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Time to objective response was defined as the time from the date of randomization to the date of the first documentation of objective response (complete response [CR] or partial response [PR]). As per Response Evaluation Criteria in Solid Tumors Version 1.1, CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: as for outcome 5
Population: Time to objective response was assessed among participants with objective response of CR or PR in the Full Analysis Set in Phase 2 of the study. Efficacy was not assessed in the Phase 1b portion of the study.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 6 | 9 | 4
weeks | 6.14 [5.29 to 6.43] | 6.29 [6.14 to 6.29] | 12.00 [6.29 to 17.29]

7. Secondary Outcome: Duration of Stable Disease Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Duration of stable disease (SD) was defined for participants whose best response is SD as the time from the date of randomization to the date of the first documentation of progressive disease. SD was defined as neither sufficient shrinkage to qualify for partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions).
Time Frame: For participants whose best response is SD as the time from date of first documentation of stable disease up to the date of first documentation of progressive disease, up to 3 years 2 months
Population: Duration of stable disease (SD) was assessed among participants with best response of SD in the Full Analysis Set in Phase 2 of the study. Efficacy was not assessed in the Phase 1b portion of the study.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 21 | 27 | 24
weeks | 25.14 [18.14 to 36.14] | 17.29 [12.86 to 24.71] | 19.57 [12.29 to 37.14]

8. Secondary Outcome: Time to Disease Progression Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Time to disease progression was defined as the time from the randomization date to the date of first objective documentation of disease progression. As per Response Evaluation Criteria in Solid Tumors Version 1.1, progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Time from date of randomization up to the date of first objective documentation of disease progression, up to 3 years 2 months
Population: Time to disease progression was assessed in the Full Analysis Set in Phase 2 of the study. Efficacy was not assessed in the Phase 1b portion of the study.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 70 | 71 | 71
weeks | 9.29 [6.14 to 16.14] | 11.14 [6.71 to 13.00] | 7.86 [6.29 to 12.14]

9. Secondary Outcome: Pharmacokinetic Parameter of Cycle 3 Patritumab Area Under the Concentration-time Curve Over the Dosing Interval 0 to τ (AUC) Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: AUC was calculated from the concentration-time data at Cycle 3 using a noncompartmental analysis (NCA) method.
Time Frame: Cycle 1: predose, end of infusion (EOI), 3 hour (h) postdose; Cycle 2: predose; Cycle 3: predose, EOI, 3 h, 6h, 24 h, 72 h, 168 h, 336 h; Cycle 4, Cycle 5, Cycle 7, and Cycle 9: predose (each cycle is 21 days)
Population: Area under the curve from 0 to tau was assessed in patients with available samples the Pharmacokinetic (PK) Analysis Set. The PK analysis sets for Phase 1b and Phase 2 were combined for the PK analyses.
Measure: Mean (Standard Deviation); unit: hour*ug/mL
Groups:
- Phase 1b and Phase 2: U31287 18 mg/kg + Erlotinib: Participants who received U3-1287 18 mg/kg intravenously (IV) every three weeks (Q3W) and Erlotinib 150 mg/day orally (PO). Phase 1b and Phase 2 PK analysis sets were combined for the PK analyses.
Arm/Group | Phase 1b and Phase 2: U31287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib
Number analyzed (Participants) | 13 | 7
hour*ug/mL | 61316.6 (29364.06) | 27713.6 (8076.02)

10. Secondary Outcome: Pharmacokinetic Parameter of Cycle 3 Patritumab Concentration End of Infusion (CEOI) and Minimum (Trough) Concentration (Cmin) Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Concentration end of infusion (CEOI) was defined as the concentration within ± 5 minutes of the end of infusion. Cmin was defined as minimum (trough) observed concentration within ± 15% of the prescribed dosing interval. Preinfusion patritumab concentrations observed within 15% of nominal time after the start of the previous infusion (ie, 21 days ± 3.15 days) were considered trough concentrations
Time Frame: as for outcome 9
Population: Concentration at end of infusion and minimum concentration were assessed in patients with available samples in the Pharmacokinetic Analysis Set. The PK analysis sets for Phase 1b and Phase 2 were combined for the PK analyses.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Phase 1b and Phase 2: U31287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib
Number analyzed (Participants) | 26 | 27
ug/mL
  CEOI | 473.67 (495.91) | 183.90 (71.82)
  Cmin: number analyzed (Participants) | 25 | 23
  Cmin | 65.86 (93.64) | 17.67 (11.48)

11. Secondary Outcome: Erlotinib Concentrations at Cycle 3 Day 1 Following U3-1287 (AMG 888) in Combination With Erlotinib
Time Frame: Cycle 3, Day 1: predose, 1 h, 2 h, 3 h, 6h, 24 h postdose (each cycle is 21 days)
Population: Erlotinib concentrations were assessed in patients with available samples in the Pharmacokinetic Analysis Set. The PK analysis sets for Phase 1b and Phase 2 were combined for the PK analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b and Phase 2: U31287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 6 | 4 | 2
ng/mL
  Predose | 837.42 (587.65) | 1547.25 (1273.15) | 1315.00 (318.20)
  1 h | 1115.50 (611.27) | 1954.00 (1249.95) | 1754.00 (1083.29)
  2 h | 1578.33 (421.83) | 1832.00 (1269.61) | 1820.00 (296.99)
  3 h | 1573.17 (481.37) | 2041.25 (1510.75) | 1855.00 (148.49)
  6 h: number analyzed (Participants) | 5 | 4 | 2
  6 h | 1902.00 (618.28) | 2362.50 (1383.51) | 1845.00 (91.92)
  24 h: number analyzed (Participants) | 6 | 3 | 2
  24 h | 1144.00 (672.69) | 2300.00 (1797.03) | 976.00 (147.08)

12. Secondary Outcome: Pharmacokinetic Parameter of Erlotinib Trough (Cmin) Concentrations From Participants Receiving 150 mg Erlotinib Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: Trough concentrations (Cmin) was defined as minimum (trough) observed concentration within ± 15% of the prescribed dosing interval. Erlotinib Cmin was predose (or for participants with at least 2 prior doses, within 15% of nominal time after postdose) plasma erlotinib concentration.
Time Frame: Cycle 1: predose, end of infusion (EOI), 3 hour (h) postdose; Cycle 2: predose; Cycle 3: predose, EOI, 3 h, 6h, 24 h, 72 h, 168 h, 336 h; Cycle 5, Cycle 7, and Cycle 9: predose (each cycle is 21 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b and Phase 2: U31287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 77 | 69 | 70
ng/mL
  Cycle 1 Day1: number analyzed (Participants) | 63 | 50 | 55
  Cycle 1 Day1 | 0 (0) | 0 (0) | 0 (0)
  Cycle 2 Day 1: number analyzed (Participants) | 18 | 14 | 19
  Cycle 2 Day 1 | 943.09 (865.13) | 1490.18 (1381.34) | 1263.47 (1328.56)
  Cycle 3 Day 1: number analyzed (Participants) | 12 | 15 | 12
  Cycle 3 Day 1 | 912.42 (785.91) | 1419.95 (911.77) | 1084.58 (851.85)
  Cycle 5 Day 1: number analyzed (Participants) | 5 | 4 | 4
  Cycle 5 Day 1 | 394.80 (256.72) | 1333.45 (1155.66) | 540.75 (307.70)
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 2 | 2
  Cycle 7 Day 1 |  | 1602.50 (1113.69) | 627.00 (19.80)
  Cycle 9 Day 1: number analyzed (Participants) | 1 | 1 | 2
  Cycle 9 Day 1 | 161.00 (NA) — Standard deviation could not be calculated on a single patient. | 1850.00 (NA) — Standard deviation could not be calculated on a single patient. | 646.50 (78.49)

13. Secondary Outcome: Treatment-Emergent Adverse Events Occurring in ≥10% of Participants Following U3-1287 (AMG 888) in Combination With Erlotinib
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that: emerged during treatment, having been absent at pretreatment; or reemerged during treatment, having been present at baseline but stopped prior to treatment; or worsened in severity since treatment relative to the pretreatment state, when the AE was continuous.
Time Frame: From the date of signing the informed consent form up to 53 days after the last dose of patritumab/placebo or up to 30 days after the last dose of erlotinib if patritumab/placebo was discontinued earlier, up to 3 years 2 months
Population: TEAEs Occurring in ≥10% of Participants Following U3-1287 (AMG 888) in Combination with Erlotinib were analyzed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: U3127 18mg/kg + Erlotinib | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
Number analyzed (Participants) | 7 | 70 | 71 | 71
Participants
  Any TEAE | 7 | 69 | 70 | 69
  Blood and Lymphatic System Disorders | 1 | 14 | 12 | 8
  Anaemia | 1 | 7 | 6 | 5
  Gastrointestinal Disorders | 7 | 59 | 58 | 38
  Abdominal distension | 1 | 0 | 0 | 1
  Abdominal pain | 1 | 9 | 9 | 3
  Abdominal pain upper | 0 | 5 | 5 | 8
  Constipation | 1 | 9 | 10 | 4
  Diarrhoea | 5 | 47 | 50 | 23
  Faecal incontinence | 1 | 0 | 0 | 0
  Gastrooesophageal reflux disease | 1 | 0 | 0 | 2
  Glossitis | 1 | 0 | 0 | 0
  Lip dry | 1 | 1 | 0 | 0
  Nausea | 3 | 26 | 17 | 14
  Oral disorder | 1 | 0 | 0 | 0
  Oral pain | 1 | 0 | 1 | 0
  Vomiting | 2 | 18 | 7 | 5
  Stomatitis | 2 | 2 | 1 | 0
  General Disorders and Administration Site Conditions | 5 | 44 | 45 | 34
  Fatigue | 4 | 18 | 22 | 13
  Gait disturbance | 1 | 1 | 0 | 0
  General physical health deterioration | 0 | 11 | 10 | 7
  Non-cardiac chest pain | 1 | 0 | 0 | 1
  Oedema peripheral | 2 | 9 | 9 | 4
  Mucosal inflammation | 2 | 1 | 5 | 1
  Pain | 1 | 0 | 0 | 0
  Temperature intolerance | 1 | 0 | 0 | 0
  Pyrexia | 0 | 8 | 6 | 4
  Asthenia | 0 | 7 | 4 | 6
  Metabolism and Nutrition Disorders | 5 | 30 | 34 | 20
  Decreased appetite | 4 | 18 | 17 | 14
  Hypokalaemia | 1 | 12 | 11 | 3
  Hypomagnesaemia | 3 | 0 | 4 | 0
  Hyponatraemia | 1 | 4 | 1 | 3
  Skin and Subcutaneous Tissue Disorders | 7 | 51 | 60 | 48
  Alopecia | 1 | 2 | 2 | 2
  Decubitus ulcer | 1 | 2 | 0 | 0
  Dermatitis acneiform | 2 | 1 | 2 | 1
  Drug eruption | 1 | 1 | 1 | 0
  Dry skin | 4 | 5 | 12 | 6
  Ecchymosis | 1 | 0 | 0 | 0
  Erythema | 1 | 1 | 0 | 0
  Onychoclasis | 1 | 0 | 1 | 1
  Pruritus | 2 | 1 | 2 | 2
  Rash | 7 | 35 | 38 | 28
  Rash generalized | 0 | 8 | 8 | 4
  Skin exfoliation | 2 | 1 | 0 | 1
  Respiratory, Thoracic, and Mediastinal Disorders | 5 | 32 | 32 | 32
  Cough | 2 | 5 | 11 | 11
  Dyspnoea | 0 | 12 | 17 | 12
  Epistaxis | 1 | 6 | 6 | 2
  Hiccups | 1 | 0 | 0 | 1
  Nasal congestion | 1 | 0 | 0 | 0
  Oropharyngeal pain | 1 | 0 | 1 | 3
  Postnasal drip | 1 | 0 | 0 | 0
  Infections and Infestations | 6 | 27 | 26 | 16
  Candidiasis | 3 | 3 | 6 | 0
  Device related infection | 1 | 1 | 0 | 0
  Fungal skin infection | 1 | 3 | 0 | 1
  Oral candidiasis | 1 | 3 | 6 | 0
  Paronychia | 0 | 8 | 5 | 1
  Tinea cruris | 1 | 0 | 0 | 0
  Urinary tract infection | 1 | 5 | 4 | 2
  Investigations | 2 | 21 | 24 | 16
  Blood creatinine increased | 1 | 1 | 2 | 0
  Blood pressure increased | 1 | 0 | 0 | 0
  Blood urea increased | 1 | 0 | 0 | 0
  Weight decreased | 1 | 10 | 16 | 8
  Cardiac Disorders | 1 | 8 | 7 | 7
  Ventricular arrhythmia | 1 | 0 | 0 | 0
  Eye disorders | 2 | 1 | 0 | 0
  Dry eye | 1 | 0 | 0 | 0
  Ocular hyperaemia | 1 | 0 | 0 | 0
  Vision blurred | 1 | 0 | 2 | 0
  Musculoskeletal and connective tissue disorders | 4 | 3 | 1 | 0
  Back pain | 2 | 6 | 3 | 4
  Flank pain | 1 | 0 | 1 | 0
  Muscular weakness | 1 | 3 | 1 | 1
  Musculoskeletal chest pain | 1 | 3 | 4 | 3
  Myalgia | 1 | 0 | 1 | 0
  Injury, poisoning and procedural complications | 4 | 6 | 9 | 2
  Contusion | 2 | 0 | 2 | 0
  Fall | 2 | 1 | 2 | 1
  Sunburn | 1 | 0 | 0 | 0
  Thermal burn | 1 | 0 | 0 | 0
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 1 | 5 | 7 | 12
  Tumour associated fever | 1 | 0 | 0 | 0
  Nervous system disorders | 5 | 4 | 2 | 3
  Ataxia | 1 | 1 | 0 | 1
  Dizziness | 1 | 0 | 1 | 0
  Dysgeusia | 2 | 1 | 2 | 1
  Headache | 2 | 2 | 3 | 2
  Hyperaesthesia | 1 | 0 | 0 | 0
  Hypoaesthesia | 1 | 0 | 0 | 0
  Paraesthesia | 1 | 0 | 1 | 2
  Peroneal nerve palsy | 1 | 0 | 0 | 0
  Presyncope | 1 | 0 | 0 | 0
  Psychiatric disorders | 2 | 11 | 12 | 12
  Anxiety | 1 | 0 | 1 | 4
  Confusional state | 1 | 0 | 0 | 1
  Depression | 1 | 3 | 3 | 3
  Insomnia | 1 | 2 | 4 | 1
  Libido decreased | 1 | 0 | 0 | 0
  Renal and urinary disorders | 4 | 7 | 2 | 2
  Haematuria | 1 | 2 | 0 | 0
  Incontinence | 1 | 0 | 1 | 0
  Nocturia | 1 | 0 | 0 | 1
  Pollakiuria | 1 | 0 | 1 | 0
  Proteinuria | 2 | 0 | 0 | 0
  Urinary hesitation | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the date of signing the informed consent form up to 53 days after the last dose of patritumab/placebo or up to 30 days after the last dose of erlotinib if patritumab/placebo was discontinued earlier, up to 3 years 2 months.
Groups:
- Phase 1b: U31287 18mg/kg + Erlotinib: Participants who received U3-1287 18 mg/kg intravenously (IV) every three weeks (Q3W) and Erlotinib 150 mg/day orally (PO).
Arm/Group | Phase 1b: U31287 18mg/kg + Erlotinib | Phase 2: U3-1287 18 mg/kg + Erlotinib | Phase 2: U3-1287 9 mg/kg + Erlotinib | Phase 2: Placebo + Erlotinib
All-Cause Mortality (participants affected / at risk) | 6/7 | 64/70 | 53/71 | 53/71
Serious Adverse Events (participants affected / at risk) | 3/7 | 35/70 | 24/71 | 24/71
Other Adverse Events (participants affected / at risk) | 7/7 | 69/70 | 70/71 | 69/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: U31287 18mg/kg + Erlotinib (N=7) | Phase 2: U3-1287 18 mg/kg + Erlotinib (N=70) | Phase 2: U3-1287 9 mg/kg + Erlotinib (N=71) | Phase 2: Placebo + Erlotinib (N=71)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 5 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3 | 3 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 4 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 2 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Panophthalmitis (Eye disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Tumor associate fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: U31287 18mg/kg + Erlotinib (N=7) | Phase 2: U3-1287 18 mg/kg + Erlotinib (N=70) | Phase 2: U3-1287 9 mg/kg + Erlotinib (N=71) | Phase 2: Placebo + Erlotinib (N=71)
Diarrhoea (Gastrointestinal disorders) | 5 | 47 | 50 | 23
Nausea (Gastrointestinal disorders) | 3 | 26 | 17 | 14
Vomiting (Gastrointestinal disorders) | 2 | 18 | 7 | 5
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 35 | 38 | 28
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 5 | 12 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 2
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Fatigue (General disorders) | 4 | 18 | 22 | 13
Mucosal inflammation (General disorders) | 2 | 1 | 5 | 1
Asthenia (General disorders) | 0 | 7 | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 4 | 18 | 17 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 12 | 11 | 3
Paronychia (Infections and infestations) | 0 | 8 | 5 | 1
Weight decreased (Investigations) | 1 | 10 | 16 | 8
Dysgeusia (Nervous system disorders) | 2 | 1 | 2 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 1 | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 7 | 6 | 5
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 9 | 9 | 3
Constipation (Gastrointestinal disorders) | 1 | 9 | 10 | 4
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 9 | 9 | 4
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 3 | 3 | 6 | 0
Device related infection (Infections and infestations) | 1 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 3 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 3 | 6 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 5 | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 1
Sunburn (Infections and infestations) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 2 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 3 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 3 | 2
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 2
Peroneal nerve palsy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 4
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 3 | 3 | 3
Insomnia (Psychiatric disorders) | 1 | 2 | 4 | 1
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 11 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 6 | 2
Hiccups (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Ecchymosis (Social circumstances) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 8 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No